CLINICAL TRIAL: NCT06032247
Title: Effect of Bilateral Versus Unilateral Lower Body Resistance Training on Musculoskeletal Outcomes in Individuals With a Previous Anterior Cruciate Ligament Reconstruction
Brief Title: Bilateral Versus Unilateral Strength Training After ACLR
Acronym: BUST
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is withdrawn due to a lack of available recruitment within the researchers' timeframe.
Sponsor: University of Kansas (Other)
Responsible Party: Principal Investigator, Christopher Cleary, MS, CPSS, CSCS, PhD Candidate, University of Kansas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150439
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Anterior Cruciate Ligament Injuries; Atrophy, Muscular; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: rehabilitation; periodization; injury risk reduction; strength training
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral strength training (Experimental): Resistance training three times per week for 8-weeks on one leg at a time per exercise.
  Interventions: Behavioral: Resistance exercise program- UL
- Bilateral strength training (Active Comparator): Resistance training three times per week for 8-weeks on both legs at a time per exercise.
  Interventions: Behavioral: Resistance exercise program- BL

INTERVENTIONS:
Behavioral: Resistance exercise program- UL — Unilateral group:
  Exercise sessions supervised by an exercise professional. Exercises will include single-leg squats, split squats, single-leg deadlifts, single-leg leg extensions, etc. Repetition range and volume (sets performed) will target strength and hypertrophy range with linear periodization utilized to ensure progression.
  Arms: Unilateral strength training
Behavioral: Resistance exercise program- BL — Bilateral group:
  Exercise sessions supervised by an exercise professional. Exercises will include double-leg squats, double-leg deadlifts, double-leg leg extensions, etc. Repetition range and volume (sets performed) will target strength and hypertrophy range with linear periodization utilized to ensure progression.
  Arms: Bilateral strength training

SUMMARY:
After rehabilitation completion, there remains large deficiencies between the operative (OP) and non-operative (NOP) limbs in lower-limb outcomes (e.g., size, strength, and function) and these deficits can persist for years. Therefore, further specialized training protocols, such as the ones in the present study, are required to determine if these deficits can be lessened. The proposed project will evaluate the effect of 8-weeks of single-leg and double-leg lower-body resistance training on musculoskeletal function in individuals with a previous anterior cruciate ligament (ACL) reconstruction (ACLR) in a randomized control trial. The study will recruit 30-40 males and females between 18-35 years of age that have undergone a previous ACLR. Participants will be randomized to either the single-leg/unilateral (UL) or double-leg/bilateral (BL) training groups. Training will occur three times per week for 8-weeks. The UL group will participate in exercises such as split squats, single-leg deadlifts, or single-leg squats. The BL group will utilize exercises such as double-leg squats, conventional deadlifts, and leg presses. One week prior to (PRE) and one week after (POST) the training program, all participants will undergo a testing battery. Musculoskeletal ultrasound will measure quadriceps and hamstrings muscle cross-sectional area (mCSA), fascicle length (FL), and pennation angle (PA) of both OP and NOP limbs. Strength will be assessed through maximal voluntary isometric contractions (MVIC) for the quadriceps and hamstrings, and one-repetition maximum tests for single-leg leg extensions, leg curls, and leg press. Lower-limb function will be assessed through single-leg and double-leg jumps on a dual force plate system for jump height, impulse, rate of force development, and peak force. Data will be analyzed via separate mixed-factorial analyses of variance for the within-subjects factor of leg (OP vs. NOP) and time (PRE vs. POST) and the between-subjects factor of biological sex (male vs. female) and group (UL vs. BL). Post-hoc analyses will include lower-order ANOVAs and t-tests as pairwise comparisons when significance is detected. Significance will be established at p≤0.05. The results of this study will assist practitioners, coaches, sport scientists, and most importantly, the athletes, in the development of post-rehabilitative strength training protocols designed to reduce between-limb discrepancies.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written and dated informed consent to participate in the study
2. Participant is 18-35 years of age, inclusive
3. Participant is in good health as determined by a health history questionnaire
4. Participant has been medically cleared to return to sport after primary ACLR in the previous two years

Exclusion Criteria:

1. Participant has a history of other lower-body related injuries in the past 6-months.
2. Participant has undergone more than one ACLR or has injured the ACL of both legs.
3. Participant has implants, hardware, devices, or other non-removable metal material in the body that would limit the accuracy of skeletal muscle size and body composition assessments within the measurement area.
4. Participant has a cardiovascular, metabolic, or neuromuscular disorder that contraindicates their ability to participate in an exercise program.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in isometric strength of the quadriceps femoris | 9-weeks
  Change in maximal voluntary isometric contraction (MVIC) peak torque (Nm) of the quadriceps from PRE (baseline) to POST
Change in muscle cross-sectional area of the quadriceps femoris | 9-weeks
  Change in absolute muscle cross-sectional area (mCSA, cm^2) of the quadriceps femoris (vastus lateralis, rectus femoris, vastus medialis) from PRE (baseline) to POST

SECONDARY OUTCOMES:
Change in muscle cross-sectional area strength of the hamstrings | 9-weeks
  Change in absolute muscle cross-sectional area (mCSA, cm^2) of the hamstrings (biceps femoris, semimembranous, semitendinosus) from PRE (baseline) to POST
Change in isometric strength of the hamstrings femoris | 9-weeks
  Change in maximal voluntary isometric contraction (MVIC) peak torque (Nm) of the hamstrings PRE (baseline) to POST
Change in jump height of both limbs | 9-weeks
  Change in jump height (cm) during countermovement jumps from PRE (baseline)
Change in jump impulse of both limbs | 9-weeks
  Change in vertical jump impulse (N/kg/s) during countermovement jumps from PRE (baseline)
Change in body composition | 9-weeks
  Change in body composition (body fat percentage (%)) assessed by bioelectrical impedance analysis (BIA) from PRE (baseline).
Change in segmental body composition | 9-weeks
  Change in segmental (legs) fat-free mass (kg) as assessed by bioelectrical impedance analysis

OTHER OUTCOMES:
Change in dynamic strength of the quadriceps and hamstrings | 9-weeks
  Change in dynamic strength (kg) of the knee extensors, knee flexors, and total thigh musculature assessed by one-repetition maximum (1-RM) testing for single-leg leg extension, single-leg leg curl, and double-leg press from PRE (baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Edwards Campus, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No